CLINICAL TRIAL: NCT01638494
Title: Calcium and Vitamin D Intakes in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Federico II University
Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 56/09
Record Dates: First submitted 2012-06-29; First posted 2012-07-11 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Hypocalcemia; Hypovitaminosis D
Keywords: 25-Hydroxyvitamin D; dietary counseling; pediatrics; allergy; bone metabolism
MeSH Terms: conditions — Hypocalcemia; Vitamin D Deficiency; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Colecalcium testing (Experimental): administration of Colecalcium
  Interventions: Dietary Supplement: Colecalcium supplement

INTERVENTIONS:
Dietary Supplement: Colecalcium supplement — Daily Ca2+ and VitD intake was determined using a previously validated written dietary questionnaire, filled by the parents with the help of a registered dietitian. Eventual assumption of Ca2+ and/or VitD supplements or fortified foods was also registered. All questionnaires were collected and analyzed using a specific software based on the Italian food composition tables (Winfood, Medimatica SRL, Martinsicuro, Teramo, Italy). All data were recorded in a specific clinical chart before statistical analysis. All subjects with less than 70% of the DRIs were invited to participate in a randomized trial aiming to investigate the efficacy of different nutritional interventions. The dietitian gave information to the parents on how to improve the consumption of foods rich in Ca2+ and VitD according to DRIs. No nutritional support products were prescribed in children enrolled in group 2.

SUMMARY:
Calcium (Ca2+) and vitamin D (VitD) play an important role in child health. Aims. The investigators evaluated the daily intake of Ca2+ and VitD in healthy children; and the efficacy of Ca2+ and VitD supplementation. Daily Ca2 + and VitD intake was evaluated in consecutive healthy children through a validated questionnaire. Subjects with a daily Ca2 + and VitD intake < 70% of dietary reference intakes (DRIs) were invited to participate in prospective randomized trial with 2 groups of nutritional intervention: group 1, dietary counseling aiming to optimize daily Ca2+ and VitD intake plus administration of a commercially available Ca2 + and VitD supplementation product (Colecalcium®, Humana, Milan, Italy); group 2, dietary counseling alone. At the enrollment (T0) and after 4 months (T1) serum VitD levels were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory healthy subjects (male and female, age range 3-17 years) consecutively observed at our Department for routine clinical examination because vaccination program were considered eligible for the study.

Exclusion criteria

* malnutrition (defined as a weight/height ratio <5° centile);
* presence of chronic systemic diseases (celiac disease, inflammatory bowel disease, food allergy, cystic fibrosis, malignancy, immunodeficiency, tuberculosis, genetic-metabolic disease, primitive bone disease, diabetes and endocrine disorder);
* and use of systemic steroids in the previous 3 months.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 184 (Actual)
Dates: Start 2008-12; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Assessed VitD intake in a population of healthy pediatric subjects and evaluate the efficacy and applicability of a nutritional intervention to optimize VitD intake. | about 1 year
  Evaluation and treatment of children with hypocalcemia and hypovitaminosis D.

SECONDARY OUTCOMES:
Assessed Ca2 intake in a population of healthy pediatric subjects and evaluate the efficacy and applicability of a nutritional intervention to optimize Ca2 intake. | about 1 year
  Evaluation and treatment of children with hypocalcemia and hypovitaminosis D.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Berni Canani, MD, PhD, Principal Investigator — Federico II University

REFERENCES:
- [Derived] Cosenza L, Pezzella V, Nocerino R, Di Costanzo M, Coruzzo A, Passariello A, Leone L, Savoia M, Del Puente A, Esposito A, Terrin G, Berni Canani R. Calcium and vitamin D intakes in children: a randomized controlled trial. BMC Pediatr. 2013 May 23;13:86. doi: 10.1186/1471-2431-13-86. PMID 23702146